CLINICAL TRIAL: NCT04912557
Title: Evaluation of the Performance of Epidural Analgesia After Major Abdominal Surgery
Acronym: PAPCAM
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/21/0160; 2021-A00926-35 (Other: IC RCB)
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Epidural Analgesia After Major Open Abdominal Surgery
Keywords: epidural analgesia; open abdominal surgery; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Open major abdominal surgery patient (predicted operative time ≥ 2 hours) with Peridural Analgesia accepted
  Interventions: Other: postoperative pain assess

INTERVENTIONS:
Other: postoperative pain assess — numerical pain scale and Metameric levels of cold insensitivity
  Other Names: numerical pain scale

SUMMARY:
Epidural analgesia is widely used for the treatment of acute postoperative pain, and currently represents the gold standard after open major abdominal surgery. However, several studies have reported a failure rate of APT of up to 30%. Its efficacy regarding pain control during coughing and mobilization is also inconsistent, with correct analgesia found in only 60% of cases in a Scandinavian multicenter cohort. Inadequate Epidural analgesia may be associated with more postoperative complications. This finding prompts a study in our institution to evaluate the performance of epidural analgesia after major open abdominal surgery.

DETAILED DESCRIPTION:
Epidural analgesia is widely used for the treatment of acute postoperative pain, and currently represents the gold standard after open major abdominal surgery. However, several studies have reported a failure rate of APT of up to 30%. Its efficacy regarding pain control during coughing and mobilization is also inconsistent, with correct analgesia found in only 60% of cases in a Scandinavian multicenter cohort. Inadequate Epidural analgesia may be associated with more postoperative complications. This finding prompts a study in our institution to evaluate the performance of epidural analgesia after major open abdominal surgery.

Epidural analgesia does not guarantee total control of acute postoperative pain after major open abdominal surgery. The performance of epidural analgesia could vary according to predisposing factors and postoperative days. Inadequate epidural analgesia could be associated with greater morbidity after open major abdominal surgery.

In order to evaluate the performance of epidural analgesia after major open abdominal surgery, a prospective observational monocentric scheme seems relevant. The evaluation will be clinical based on questioning and a brief medical examination during the early postoperative phase of the operated patients.

ELIGIBILITY:
Inclusion Criteria:

* Major abdominal surgery patient operated by laparotomy (predicted operative time ≥ 2 hours)
* epidural analgesia accepted

Exclusion Criteria:

* Minor or protected patient
* Patients under guardianship, curatorship or safeguard of justice
* Pregnant or breastfeeding woman
* Contraindication or refusal of epidural analgesia
* Failure of the initial placement of the epidural catheter
* Major intraoperative complication requiring continued postoperative sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients with major abdominal surgery operated by laparotomy
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2021-12-11 (Actual); Study Completion 2021-12-11 (Actual)

PRIMARY OUTCOMES:
Insufficient epidural analgesia | day 5
  Insufficient epidural analgesia will be defined by the presence of pain assessed by numerical scale > 3/10 at rest OR on coughing OR on mobilization.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume PORTA-BONETE, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No